CLINICAL TRIAL: NCT03618875
Title: Reduction of Post Intravitreal Injection Bleeding and Pain by Ice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: icepreventpain
Record Dates: First submitted 2017-11-26; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2016-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ice (Active Comparator): Patients were randomly assigned to receive an ice 5 minutes prior the IViT
  Interventions: Other: ice pack
- placebo (Placebo Comparator): Patients were randomly assigned to a room temperature patch (placebo) 5 minutes prior the IViT
  Interventions: Other: room temperature pack

INTERVENTIONS:
Other: ice pack — ice pack was placed on eyelid 5 minutes prior to IVIT
  Arms: ice
Other: room temperature pack — room temperature pack was placed on eyelid 5 minutes prior to IVIT
  Arms: placebo

SUMMARY:
Intravitreal injections are an efficient method for delivering intraocular therapeutic agents in numerous ophthalmologic diseases. However, side effects, such as pain and subconjunctival hemorrhage remain a major concern.

Prevention or alleviation of those side effects might shorten the healing duration and improve patients' quality of life.

DETAILED DESCRIPTION:
cooling the eye using ice patched prior to Intravitreal injections may ameliorated pain and subconjunctival hemorrhage incidences.

ELIGIBILITY:
Inclusion Criteria:

patients receiving intravitreal injection

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-25 (Actual)

PRIMARY OUTCOMES:
pain | change between VAS pain score at baseline and 10 minutes
  Visual Analogue Scale (VAS) is a Likert-type scale (1-10). The VAS is a reliable tool in evaluating and quantifying ocular discomfort

SECONDARY OUTCOMES:
size of subconjunctival hemorrhage | change between subconjunctival hemorrhage at baseline and 10 minutes
  subconjunctival hemorrhage in mm

CONTACTS AND LOCATIONS:
Locations (1):
- The E.Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No
no plan